CLINICAL TRIAL: NCT05334446
Title: The Effect on Treatment Compliance and Self-Care Management in Patients With Hypertension
Brief Title: The Effect ''of Follow-up With the Mobile Application'' on Treatment Compliance in Patients With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Alev Yıldırım Keskin, Assistant Professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021/19; 2021/484 (Registry Identifier: Mobile Application in Patients with Hypertension)
Record Dates: First submitted 2022-03-14; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Hypertension
Keywords: Hypertension; Mobile Application; Treatment Compliance; Self Care Management
MeSH Terms: conditions — Hypertension; Patient Compliance

STUDY DESIGN:
Intervention Model Description: The Effect ''of Follow-up With the Mobile Application'' on Treatment Compliance with the intervention group.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Effect ''of Follow-up with the Mobile Application'' in Patients with Hypertension (Experimental): Intervention Group:mobile application for 4 weeks; This is the training group in which individual motivational messages will be sent to the mobile phones every week for compliance with the diet, exercise and drug therapy of the patients, and the weekly average of blood pressure follow-ups is monitored over the system.
  Interventions: Behavioral: The Effect of the Mobile Application
- The Effect ''of Follow-up with the Mobile Application'' in Hypertension control group (No Intervention): It is the control group whose routine outpatient follow-up will continue and no training is given

INTERVENTIONS:
Behavioral: The Effect of the Mobile Application — This study was planned to determine the "Effect of Mobile Application Use on Treatment Adherence and Self-Care Management in Patients with Hypertension". The study was designed to improve individuals' knowledge about the disease, regular drug use, diet compliance, physical activity level, quitting smoking and alcohol if using, and weight control.
  Arms: The Effect ''of Follow-up with the Mobile Application'' in Patients with Hypertension

SUMMARY:
Hypertension is an important disease that generally affects the adult population, is increasing rapidly in our country and in the world, and threatens public health due to its complications. In our country, the rate of blood pressure control in patients receiving antihypertensive treatment is 53.9%. One of the factors that play a role in not exceeding this rate is the patient's non-compliance with treatment.

Hypertension management has two main building blocks. These are: lifestyle improvement and drug therapy. According to the data of the World Health Organization, the rate of compliance with treatment in chronic diseases in developing countries is around 50%. Morbidity and mortality are directly related to the use of drugs in patients with hypertension, and the control of hypertension is possible with the patient's compliance with the treatment. Among the reasons for non-compliance with treatment; The side effects of drugs, the patient's insecurity about the effectiveness and benefit of the treatment, lack of motivation, the absence of disturbing physical symptoms in some patients, lack of knowledge about drug therapy and diet regimens, miscommunication between the patient and the physician, the complexity of the treatment, and insufficient participation in the follow-up of the patient can be counted. It is important to support and follow-up the hypertensive individual in order to develop their self-care skills and to adapt and maintain their lifestyle changes and drug treatment to keep their blood pressure under control.

The use of mobile health services is becoming more and more popular in the self-management of chronic diseases such as hypertension. Due to the rapid adoption of smartphone technologies, mobile phones are now attracting the attention of individuals with chronic diseases and increasing their usability, thanks to their entertaining use as well as monitoring patient data, providing personalized self-management, benefiting from social effects.

This study was planned to determine the "Effect of Mobile Application Use on Treatment Adherence and Self-Care Management in Patients with Hypertension". The study was designed to improve individuals' knowledge about the disease, regular drug use, diet compliance, physical activity level, quitting smoking and alcohol if using, and weight control.

DETAILED DESCRIPTION:
This research was planned as a randomized controlled study in the pre-test post-test evaluation order before and after the mobile application in order to determine the "Effect of Mobile Application Use on Treatment Adherence and Self-Care Management in Patients with Hypertension".

The research was carried out between 22.11.2021-03.01.2022. It is planned to be conducted with patients who applied to the Cardiology Polyclinic of City Hospital and who were diagnosed with essential hypertension at least 1 year ago and met the research criteria.

The sample of the study, on the other hand, will consist of patients aged 18 and over, who were diagnosed at least 1 year ago, who were diagnosed with hypertension, who applied to the hypertension outpatient clinic, who were treated with antihypertensive drugs, who met the inclusion criteria of the study, and who volunteered to participate in the study. G-power program was used for power calculation of the study. Accordingly, it was calculated that at least 30 participants in each group were required for a difference of at least 5% between the control and intervention groups to be significant at the 95% confidence interval for 80% power. When the 10% loss that may occur during the follow-up of the patients is added to this number, it was planned to include at least 33 participants for both groups.

Sample selection in this study; Randomization will be performed by a person who was not involved in the study in the computer environment. Those with odd number of patient registration numbers will be Group 1: Intervention (Training Group), those with even number of patient registration numbers will be Group 2: Control Group.

Group 1: To be followed by the researchers for 4 weeks with a mobile application; This is the training group in which individual motivational messages will be sent to the mobile phones every week for compliance with the diet, exercise and drug therapy of the patients, and the weekly average of blood pressure follow-ups will be monitored over the system.

Group 2: It is the control group whose routine outpatient follow-up will continue and no training is given.

Data Collection Tools to be Used in the Study: Data collection form will be collected with "Hill-Bone Hypertension Treatment Adherence Scale", "Hypertension Self-Care Profile Scale".

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study,
* Being followed in the outpatient clinic with the diagnosis of hypertension for the last 1 year,
* Using antihypertensive medication
* Being a smart mobile phone user,
* 18 years of age and over
* Not having any communication problems such as seeing or hearing,
* Ability to read and write

Exclusion Criteria:

* Those who lost their lives during the research,
* Those who want to leave the research voluntarily at any stage of the research,
* Patients who fill in the forms incompletely and have missing data will be excluded from the study.
* Being illiterate
* Having communication problems such as seeing and hearing,
* Not being willing to participate in the study,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Blood pressure value | 6 weeks
  The average blood pressure values of the patients will be taken at the end of 24 hours by attaching a blood pressure holter.
Hypertension Self-Care Profile Scale | 6 weeks
  Motivation of patients; It is a 20-item Likert-type scale evaluating not important=1, somewhat important=2, important=3, very important=4. The scale results in a score between 20 and 80. A higher score indicates better self-care of a patient with hypertension.
Hill-Bone Hypertension Treatment Adherence Scale | 6 weeks
  The scale consists of 14 questions of 4-point Likert type. The answers include (0) "Never", (1) "Sometimes", (2) "Often" and (3) "Always". The scale total score ranges from 0 to 42. The higher the score, the lower the fit.

CONTACTS AND LOCATIONS:
Overall Officials: Alev YILDIRIM KESKİN, Asst. Prof, Principal Investigator — Selcuk University/ School of Health, KONYA, TURKEY
Locations (1):
- Alev YILDIRIM KESKİN, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marquez Contreras E, Marquez Rivero S, Rodriguez Garcia E, Lopez-Garcia-Ramos L, Carlos Pastoriza Vilas J, Baldonedo Suarez A, Gracia Diez C, Gil Guillen V, Martell Claros N; Compliance Group of Spanish Society of Hypertension (SEH-LELHA). Specific hypertension smartphone application to improve medication adherence in hypertension: a cluster-randomized trial. Curr Med Res Opin. 2019 Jan;35(1):167-173. doi: 10.1080/03007995.2018.1549026. Epub 2018 Dec 5. PMID 30431384
- [Background] Kang H, Park HA. Development of Hypertension Management Mobile Application based on Clinical Practice Guidelines. Stud Health Technol Inform. 2015;210:602-6. PMID 25991219
- [Background] Hallberg I, Ranerup A, Kjellgren K. Supporting the self-management of hypertension: Patients' experiences of using a mobile phone-based system. J Hum Hypertens. 2016 Feb;30(2):141-6. doi: 10.1038/jhh.2015.37. Epub 2015 Apr 23. PMID 25903164
- [Background] Bengtsson U, Kjellgren K, Hallberg I, Lindwall M, Taft C. Improved Blood Pressure Control Using an Interactive Mobile Phone Support System. J Clin Hypertens (Greenwich). 2016 Feb;18(2):101-8. doi: 10.1111/jch.12682. Epub 2015 Oct 12. PMID 26456490
- [Background] Cutrona SL, Choudhry NK, Fischer MA, Servi A, Liberman JN, Brennan TA, Shrank WH. Modes of delivery for interventions to improve cardiovascular medication adherence. Am J Manag Care. 2010;16(12):929-42. PMID 21348564
- [Background] Bengtsson U, Kjellgren K, Hallberg I, Lundin M, Makitalo A. Patient contributions during primary care consultations for hypertension after self-reporting via a mobile phone self-management support system. Scand J Prim Health Care. 2018 Mar;36(1):70-79. doi: 10.1080/02813432.2018.1426144. Epub 2018 Jan 18. PMID 29343156
- [Derived] Yildirim Keskin A, Ozpancar Solpan N, Degirmenci H. The Effect of Mobile Application Follow-Up on Treatment Compliance and Self-Care Management in Patients With Hypertension: Randomized Controlled Trial. Public Health Nurs. 2025 Jan-Feb;42(1):275-285. doi: 10.1111/phn.13476. Epub 2024 Nov 4. PMID 39492655